CLINICAL TRIAL: NCT05026086
Title: Effects of Isometric Exercises With and Without Pressure Biofeedback on Cervical Pain and Muscle Strength in Computer Users With Cervical Spine Overload
Brief Title: Isometric Exercises With and Without Pressure Biofeedback in Computer Users With Cervical Spine Overload
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/21/0115
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Pain, Neck
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biofeedback (Experimental): 10 patients will be treated with isometric exercises and pressure biofeedback.
  Interventions: Other: pressure biofeedback
- isometric exercises (Active Comparator): 10 patients will be treated with isometric exercises without pressure biofeedback.
  Interventions: Other: isometric exercises

INTERVENTIONS:
Other: pressure biofeedback — 10 patients will be treated with isometric exercises and pressure biofeedback.
  Arms: biofeedback
Other: isometric exercises — 10 patients will be treated with isometric exercises
  Arms: isometric exercises

SUMMARY:
Neck pain is defined as the pain experienced from the base of the skull or occiput to the upper part of the back and extending laterally to the outer and superior bounds of the shoulder blade. Office work is a kind of job that demands sitting for prolonged time requiring the use of computer. These two factors are mainly responsible for overloading of the spine. Neck pain and computer users are clearly connected due to extended periods of sitting in a certain position with no breaks to stretch the neck muscles. Prolonged computer use with neck bent forward will cause the anterior neck muscles to gradually get shorter and tighter, while the muscles in the back of neck will grow longer and weaker. These changes will lead to development of neck pain. Neck problem also accounts for a large proportion of occupational illness and disability. Neck pain is common among computer workers in our country and contributes importantly to the demand for medical services and the economic burden of absence from work due to sickness.

The main purpose of this randomized clinical trial will be to find out the effects of Isometric exercises with and without Pressure Biofeedback Unit on Cervical pain and Muscle strength in Computer users with cervical spine overload. Patients will be recruited in the study by convenient sampling technique after that will be allocated to groups by simple random assignment with an inclusion criteria having chronic neck pain for more than 3 months, current pain level ranging greater than 3 on NPRS, patient with minimum and moderate disability and male and female computer users with age 25 to 40 years with cervical pain. Patients with history of cervical trauma, postural deformity, spinal cord deformity, current pregnancy and significant neurological deficits were excluded.

Numeric Pain Rating Scale (NPRS) and Neck Disability Index (NDI) will be used to measure before and after treatment session. Treatment will be given to both groups for 4 weeks and each group will receive 3 sessions per week. After collecting the data it will entered and analysed using Statistical Package for the Social Sciences (SPSS) version 25. Data will be assessed by using parametric/ non parametric test after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20-40 years among male and female with cervical pain
* Having chronic pain for more than 3 months.
* Current pain level ranging greater than 3 on NPRS
* Patients with minimum and moderate disability based on NDI

Exclusion Criteria:

* History of cervical trauma
* Postural deformity
* Spinal cord deformity ( scoliosis, kyphosis, lordosis)
* Current pregnancy
* Significant neurological deficits ( cervical radiculopathy, cervical spondylosis)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
pain of patient | 4 weeks
  NPRS The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
function | 4 weeks
  Neck Disability index (NDI) Item scores range from 0 to 5, and the total score is a total of the item scores (possible range 0 (no pain) - 100 (maximal pain)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Muhammad Hahim, Lahore, Ppunjab, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen SP, Hooten WM. Advances in the diagnosis and management of neck pain. BMJ. 2017 Aug 14;358:j3221. doi: 10.1136/bmj.j3221. PMID 28807894
- [Background] Barrett JM, McKinnon C, Callaghan JP. Cervical spine joint loading with neck flexion. Ergonomics. 2020 Jan;63(1):101-108. doi: 10.1080/00140139.2019.1677944. Epub 2019 Oct 15. PMID 31594480
- [Background] Genebra CVDS, Maciel NM, Bento TPF, Simeao SFAP, Vitta A. Prevalence and factors associated with neck pain: a population-based study. Braz J Phys Ther. 2017 Jul-Aug;21(4):274-280. doi: 10.1016/j.bjpt.2017.05.005. Epub 2017 May 20. PMID 28602744
- [Background] Khan R, Surti A, Rehman R, Ali U. Knowledge and practices of ergonomics in computer users. J Pak Med Assoc. 2012 Mar;62(3):213-7. PMID 22764450